CLINICAL TRIAL: NCT05718921
Title: A Randomized, Double-blind, Placebo-controlled Single and Multiple Dose Phase I Clinical Trial to Investigate the Safety, Tolerability and Pharmacokinetics of Topical Ointment YR001 in Adult Healthy Volunteers
Brief Title: A Safety, Tolerability and Pharmacokinetics Study of Topical Ointment YR001 in Adult Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hangzhou Yirui Pharmaceutical Technology Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: YR001-A01
Record Dates: First submitted 2023-01-30; First posted 2023-02-08 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Atopic Dermatitis; Psoriasis
MeSH Terms: conditions — Dermatitis, Atopic; Psoriasis

STUDY DESIGN:
Intervention Model Description: This study includes two sequential parts of single dose and multiple dose with placebo control
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (12):
- Part A, Active dose A and Low body surface area (Experimental): The intervention is YR001 Dose A on low body surface area, low dose YR001 for single topical administration
  Interventions: Drug: YR001 Dose A on low body surface area
- Part A, Active dose A and Middle body surface area (Experimental): The intervention is YR001 Dose A on middle body surface area, low dose for single topical administration
  Interventions: Drug: YR001 Dose A on middle body surface area
- Part A, Active dose A and High body surface area (Experimental): The intervention is YR001 Dose A on high body surface area, low dose for single topical administration
  Interventions: Drug: YR001 Dose A on high body surface area
- Part A, Active dose B and Low body surface area (Experimental): The intervention is YR001 Dose B on low body surface area, high dose YR001 for single topical administration
  Interventions: Drug: YR001 Dose B on low body surface area
- Part A, Active dose B and Middle body surface area (Experimental): The intervention is YR001 Dose B on middle body surface area, high dose YR001 for single topical administration
  Interventions: Drug: YR001 Dose B on middle body surface area
- Part A, Active dose B and High body surface area (Experimental): The intervention is YR001 Dose B on high body surface area, high dose YR001 for single topical administration
  Interventions: Drug: YR001 Dose B on high body surface area
- Part A, Placebo and Low body surface area (Placebo Comparator): The intervention is Placebo on low body surface area, Placebo for single topical administration
  Interventions: Drug: Placebo on low body surface area
- Part A, Placebo and Middle body surface area (Placebo Comparator): The intervention is Placebo on middle body surface area, Placebo for single topical administration
  Interventions: Drug: Placebo on middle body surface area
- Part A, Placebo and High body surface area (Placebo Comparator): The intervention is Placebo on high body surface area, Placebo for single topical administration
  Interventions: Drug: Placebo on high body surface area
- Part B, Active dose A and High body surface area (Experimental): The intervention is YR001 Dose A on high body surface area twice daily, low dose YR001 for multiple topical administration
  Interventions: Drug: YR001 Dose A on high body surface area twice daily
- Part B, Active dose B and High body surface area (Experimental): The intervention is YR001 Dose B on high body surface area twice daily, high dose YR001 for multiple topical administration
  Interventions: Drug: YR001 Dose B on high body surface area twice daily
- Part B, Placebo and High body surface area (Placebo Comparator): The intervention is Placebo on high body surface area twice daily, Placebo for multiple topical administration
  Interventions: Drug: Placebo on high body surface area twice daily

INTERVENTIONS:
Drug: YR001 Dose A on low body surface area — Part A: Single topical dose
  Arms: Part A, Active dose A and Low body surface area
Drug: YR001 Dose A on middle body surface area — Part A: Single topical dose
  Arms: Part A, Active dose A and Middle body surface area
Drug: YR001 Dose A on high body surface area — Part A: Single topical dose
  Arms: Part A, Active dose A and High body surface area
Drug: YR001 Dose B on low body surface area — Part A: Single topical dose
  Arms: Part A, Active dose B and Low body surface area
Drug: YR001 Dose B on middle body surface area — Part A: Single topical dose
  Arms: Part A, Active dose B and Middle body surface area
Drug: YR001 Dose B on high body surface area — Part A: Single topical dose
  Arms: Part A, Active dose B and High body surface area
Drug: Placebo on low body surface area — Part A: Single topical dose
  Arms: Part A, Placebo and Low body surface area
Drug: Placebo on middle body surface area — Part A: Single topical dose
  Arms: Part A, Placebo and Middle body surface area
Drug: Placebo on high body surface area — Part A: Single topical dose
  Arms: Part A, Placebo and High body surface area
Drug: YR001 Dose A on high body surface area twice daily — Part B: Multiple topical dose
  Arms: Part B, Active dose A and High body surface area
Drug: YR001 Dose B on high body surface area twice daily — Part B: Multiple topical dose
  Arms: Part B, Active dose B and High body surface area
Drug: Placebo on high body surface area twice daily — Part B: Multiple topical dose
  Arms: Part B, Placebo and High body surface area

SUMMARY:
This study is to evaluate the safety, tolerability, and pharmacokinetics of YR001 topical ointment in healthy adult subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent obtained from the subject
2. Male or female subject is aged between 18 and 65 years
3. Subject has a weight of at least 50 kg and a body mass index (BMI) between 18.0 and 30.0 kg/m2
4. Free from any clinically relevant illness or disease incl. skin disorder that may adversely affect the safety of the subject or the integrity of the study

Exclusion Criteria:

1. Presence or history of a clinically significant medical condition or other condition that might interfere with the safety, tolerability and PK assessment of ointment YR001, or place the subject at an unacceptable risk as a subject in this study.
2. Pregnant or lactating women.
3. Any skin tattoo, scar, cuts, bruises, or other skin damage, including excessive UV exposure, at the possible IP application sites.
4. Have concomitant skin disease or infection (e.g., acne, impetigo) or presence of skin comorbidities in the skin areas to be dosed that may interfere with study assessments and treatment response.
5. Have active infectious disease.
6. Subjects treated with another investigational drug, biological agent, or device
7. Participation in another interventional clinical trial before entering, or during the trial, or previous participation in this clinical trial.
8. Evidence of clinically important cardiac conduction abnormalities at screening as judged by ECG.
9. Active untreated mental or psychiatric disorder.
10. Any major surgery within 6 months of screening.
11. Malignancy within 5 years, except for basal or squamous cell carcinoma of the skin or carcinoma in situ of the cervix that has been successfully treated.

13. Drug or alcohol abuse history.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2023-04-08 (Actual); Primary Completion 2023-08-14 (Actual); Study Completion 2023-12-14 (Actual)

PRIMARY OUTCOMES:
Part A: Safety and Maximum Tolerate Dose (MTD) | day 0 to day 8
  Incidence of treatment related AEs (TRAEs) and local skin tolerance
Part B: Safety and Maximum Tolerate Dose (MTD) | day 0 to day 22
  Incidence of treatment related AEs (TRAEs) and local skin tolerance

SECONDARY OUTCOMES:
Part A: all treatment-emergent AEs | day 0 to day 8
  Number, severity, causality, and outcome of all treatment-emergent AEs (TEAEs)
Part B: all treatment-emergent AEs | day 0 to day 22
  Number, severity, causality, and outcome of all treatment-emergent AEs (TEAEs)

CONTACTS AND LOCATIONS:
Overall Officials: Stacy Smith, Dr. MD, Study Director — Encinitas, California USA
Locations (1):
- California Dermatology & Clinical Research Institute, Encinitas, California, United States

IPD SHARING:
Plan to Share IPD: No